CLINICAL TRIAL: NCT07302867
Title: Neuromodulation in Treatment Resistant Essential Tremor in Early Habituation - Investigating Low and High Frequencies / Waveform Shaping / Pulse and Bursts / Combination Therapy in Deep Brain Stimulation Utilizing the Boston Scientific® Chronos™ Software
Brief Title: Neuromodulation Strategies for Treatment-Resistant Essential Tremor Using Chronos™ DBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Christopher Honey, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H25-03800
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation; Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Appointments and Schedules

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-group assignment interventional study. All enrolled participants undergo a structured trial of six experimental DBS stimulation paradigms delivered through Chronos™ software. Participants are then randomized to one stimulation program for at-home use. There is no comparison group; all participants receive active intervention. Follow-up occurs at 4 weeks, 3 months, and optionally at 1 year to assess tremor response, durability of benefit, and safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Experimental Arm (Experimental): All participants will test six different experimental DBS stimulation programs in the clinic using Chronos™ software. After trying all six programs, each participant will be randomly assigned to one of the six stimulation patterns to use at home for the study period. There is no control or placebo group; all participants receive an active DBS programming intervention.
  Interventions: Other: Continuous; Other: Continuous + High Frequency Cycling; Other: High Frequency; Other: Microburst; Other: Scheduling; Other: Cycling

INTERVENTIONS:
Other: Continuous — DBS setting: 185 Hz, 60 µs pulse width, optimized amplitude
Other: Continuous + High Frequency Cycling — DBS setting: Alternates 30s at 185 Hz and 30s at 1000 Hz
Other: High Frequency — DBS setting: 1000 Hz continuous, 60 µs, optimized amplitude
Other: Microburst — DBS setting: 900 Hz intraburst, 80 Hz interburst, 6 pulses per packet
Other: Scheduling — DBS setting: Two or three effective programs on alternating schedules
Other: Cycling — DBS setting: 30s on / 5s off cycle without ramp, subthreshold stimulation

SUMMARY:
The goal of this observational study is to learn whether a new way of programming Deep Brain Stimulation (DBS) can improve and maintain tremor control in adults with essential tremor (ET) who stopped responding to standard DBS therapy.

The main questions it aims to answer are:

* 1. Can advanced DBS settings, using varied stimulation patterns, frequencies, and pulses, restore tremor control in people with ET who lost benefit from standard Ventral Intermedius Deep Brain Stimulation (VIM-DBS)?
* 2. Do these advanced settings provide more stable, longer-lasting tremor improvement over time?

Researchers will compare six different stimulation settings to see if any of them can improve tremor symptoms when standard DBS programming no longer works.

Participants will:

* Complete a clinic visit where they try six different DBS stimulation settings using specialized Chronos software.
* Be randomly assigned to one of these settings to use at home.
* Receive a follow-up phone call at 4 weeks to check on symptoms and device use.
* Return to the clinic at 3 months for a full tremor evaluation.
* Have the option to return for an additional follow-up visit at 1 year.

This study will include 5 participants with essential tremor who previously lost benefit quickly after receiving standard VIM-DBS treatment.

DETAILED DESCRIPTION:
* Purpose: To test whether new DBS programming patterns can restore and sustain tremor control in essential tremor (ET) patients who lose benefit quickly after standard Vim-DBS.
* Hypothesis: Novel stimulation paradigms - like high-frequency, microburst, cycling, and scheduling - can overcome early habituation and provide lasting tremor improvement.
* Justification: Some ET patients experience rapid loss of benefit despite correct DBS placement. Standard programming does not help them, creating a disabling condition. Advanced programming may offer a safe, non-surgical solution.
* Objectives:
* 1. Determine if Chronos™ software programs maintain tremor improvement beyond one month.
* 2. Assess safety, tolerability, and identify the most effective stimulation parameters.
* Research Design: Prospective, single-center cohort study of 5 early-habituating ET patients. Patients trial six stimulation paradigms in clinic, then are randomized to one program for home use. Follow-up occurs at 4 weeks, 3 months, and optionally 1 year.
* Statistical Analysis: Descriptive statistics due to small sample size. Outcomes include tremor ratings, patient-reported benefit, and recurrence of habituation.

ELIGIBILITY:
Inclusion Criteria:

* Adults with essential tremor who have undergone standard Vim-DBS surgery
* Demonstrated rapid (early) habituation to standard programming.
* Ability to provide informed consent and attend follow-up visits.

Exclusion Criteria:

* Inability to attend programming visits.
* Cognitive or language impairment precluding consent.
* Other neurological conditions confounding tremor assessment.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
The Fahn-Tolosa-Marín Tremor Rating Scale (FTM-TRS) | 3-Month post programming

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No